CLINICAL TRIAL: NCT04749329
Title: Randomized Double-blind Study on the Use of Resorbable Prosthetic Mesh "Ante Rectus" as a Prevention of Parastomal Hernia in Patients Undergoing Terminal Colostomy
Brief Title: Use of Resorbable Prosthetic Mesh "Ante Rectus" as Prevention of Parastomal Hernia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Sanitaria Locale Napoli 2 Nord (Other)
Responsible Party: Principal Investigator, Francesco Pizza, Head of Bariatric Unit, Azienda Sanitaria Locale Napoli 2 Nord
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 212128
Record Dates: First submitted 2021-02-07; First posted 2021-02-11 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Parastomal Hernia

STUDY DESIGN:
Intervention Model Description: This study is a Binary outcome superiority trial. The sample size was calculated by Sealed Envelope Ltd. 2012. The calculation was based on the evaluation of PH rate at 3, 6, 12 and 24 months postoperatively in patients undergoing colostomy. In literature same trials reported a decrease in the incidence of PH in the mesh groups versus suture alone (xx). Therefore, we hypothesized a decrease of PH between Control and Mesh group of 25% (from 35 % to 10%). It was estimated that 49 subjects per group would be required to detect an absolute improvement of 25% (35% vs 10%) in the primary outcome between the two groups, with two-tailed α of 0.05 (2-sided 5% significance level) and a power of 80%. Data analysis was conducted according to an intention-to-treat approach. Loss to follow-up was estimated in about 10% of included patients. Therefore, a total of 110 patients (55 for each group) were included in the study.
Who Masked: Participant, Investigator
Masking Description: Patients were randomized in two groups (Control Group, without mesh; Mesh Group, receiving Bio-A mesh supported colostomy in an ante rectus fashion). Participants were randomly allocated to one of the two groups using computer-generated permuted blocks (www.randomization.com), just before colostomy fashion. For each patient, an identification number was generated. This latter was utilized during all the follow-up period guarantying the blinding process. Patients, care providers, staff collecting data and those assessing the endpoints, in fact, we're all blinded to group allocation. Because the blinding of the operating surgeons was not feasible, they were not involved in the
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): no mesh was used for end colostomy fashions
- Mesh Group (Experimental): Mesh of Bio A was used for end colostomy fashions
  Interventions: Device: Mesh Group

INTERVENTIONS:
Device: Mesh Group — All MG patients underwent the procedure with ante rectus positioned prophylactic mesh according to the following standardized technique. A BIO-A circular-shaped mesh measuring 8X10 cm in diameter is prepared with an internal 2 cm hole to let the bowel pass.
  An at least 8x8 cm space is created between the anterior rectus sheath and the rectus abdominis muscle and, then, the mesh is positioned. The bowel is passed through the rectus muscle via the circular incision in the middle of the mesh. Single absorbable monofilament sutures anchored the mesh laterally in the ante rectus pocket, while medially the mesh is fixed with four stitches to the colon and to both the anterior rectal sheet. The stoma is attached to the skin similarly to CG patients.
  Arms: Mesh Group

SUMMARY:
The aim of this study was to assess feasibility, potential benefits and safety of a prophylactic biosynthetic mesh placed at the time of colostomy.

DETAILED DESCRIPTION:
Several surgical scenarios include colon diversion as part of their management. Among them, the most frequent conditions requiring colostomy are abdominal malignancies, large bowel diverticulitis, Inflammatory Bowel Disease, bowel obstruction or perforation and postoperative complications such as anastomotic leakage. Colostomy related morbidity includes retraction, infection, prolapse, skin problems and parastomal hernia. Parastomal Hernia is a quite common late complication, with a clinical rate up to 55%, reaching 80% when assessed by Computer Tomography. Although Parastomal Hernia is often asymptomatic, significant morbidity exists, including pain, intermittent obstruction, stoma leakage, skin irritation and pouching, often reducing patients' Quality of Life. Several surgical options are available for Parastomal Hernia repair, many of them supporting the use of mesh to strengthen the fascia. However, results are often disappointing with quite high recurrence rates, rising up to 33%, even with the use of a mesh. Several studies have been published, testing effectiveness and safety of a prophylactic mesh in vertical laparotomy closure to prevent incisional hernia.

The aim of this study was to assess feasibility, potential benefits and safety of a prophylactic biosynthetic mesh placed at the time of colostomy.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* endo colostomy
* Informed consent

Exclusion Criteria:

* age < 18 years;
* life expectancy < 24 months (as estimated by the operating surgeon)
* pregnancy
* immunosuppressant therapy within 2 weeks before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Parastomal Hernia at clinical control. | 3 months
  Detect of paratoia hernia
Rate of Parastomal Hernia at clinical control. | 6 months
  Detect of paratoia hernia
Rate of Parastomal Hernia at clinical control. | 12 months
  Detect of paratoia hernia
Rate of Parastomal Hernia at clinical control. | 24 months
  Detect of paratoia hernia

SECONDARY OUTCOMES:
Rate of Parastomal Hernia at tomography observation. | 3 months follow-up
  detect of parastomal hernia
Rate of Parastomal Hernia at tomography observation. | 6 months follow-up
  detect of parastomal hernia
Rate of Parastomal Hernia at tomography observation. | 12 months follow-up
  detect of parastomal hernia
Rate of Parastomal Hernia at tomography observation. | 24 months follow-up
  detect of parastomal hernia
Number of patients affected by Superficial surgical site infections | Within 30 days postoperatively
  Superficial infections according to Clavien-Dindo criteria
Number of patients affected by Deep surgical site infections | Within 30 days postoperatively
  Deep surgical site infections according to Clavien-Dindo criteria

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Pizza, Md, PhD, Principal Investigator — Azienda Sanitaria Locale Napoli 2 Nord
Locations (2):
- Italy (2):
  - Aslnapoli2Nord, Naples
  - francesco Pizza, Naples

IPD SHARING:
Plan to Share IPD: No